CLINICAL TRIAL: NCT05475561
Title: Comparison of Erector Spinae Plane Block and Pecto-Intercostal Facial Plane Block For Enhanced Recovery After Sternotomy in Adult Cardiac Surgery
Brief Title: Comparison of Erector Spinae Block and Pecto-Intercostal Facial Block For Enhanced Recovery in Adult Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0305600
Record Dates: First submitted 2022-07-07; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-05

CONDITIONS: Cardiac Septal Defects With Coarctation of the Aorta; Mitral Regurgitation
MeSH Terms: conditions — Cardiac Septal Defects with Coarctation of the Aorta; Mitral Valve Insufficiency | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (P) (Active Comparator)
  Interventions: Procedure: Ultrasound guided Pecto-intercostal- fascial plane block; Drug: Bupivacain
- Group (E) (Active Comparator)
  Interventions: Procedure: Ultrasound guided erector spinae plane block; Drug: Bupivacain

INTERVENTIONS:
Procedure: Ultrasound guided Pecto-intercostal- fascial plane block — The probe of the ultrasound will be placed at 2 cm lateral to the lateral sternal border at 5th and 6th rib. On the surface plane subcutaneous tissue is identified, while Pectoralis major muscle, Intercostal muscles and ribs are seen in intermediate plane and lung along with pleura are identified in deep plane. A 22-gauge, 80-mm short bevel echogenic needle is used and advanced in in-plane manner, in a caudal-to-cranial direction, until the tip of the needle is located in the fascial plane between the pectoralis major and internal intercostal muscle, where the local anesthetic will be injected.
  Arms: Group (P)
Procedure: Ultrasound guided erector spinae plane block — A high-frequency linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T6 spinous process corresponding to the T5 transverse process. Three muscles trapezius (uppermost), rhomboids major (middle), and erector spinae (lowermost) will be identified superior to the hyperechoic transverse process.Local infiltration with 2% of lignocaine at the site of needle insertion will be done. Using in-plane approach a 22 G short bevel needle will be inserted in caudal-cephalad direction, until the tip is deep to erector spinae muscle, as evidenced by visible hydro dissection below the muscle plane. A 20 ml of 0.25% plain bupivacaine will be injected on each side.
  Arms: Group (E)
Drug: Bupivacain — local anesthetic

SUMMARY:
The current study is designed to compare the perioperative analgesic efficacy of Erector spinae plane block (ESPB) and Pecto-intercostal-fascial plane block (PIFB) in adults undergoing cardiac surgery via median sternotomy.

The primary outcome measure will be the analgesic effectiveness of both blocks in median sternotomy pain, while the secondary outcome measures will be time to extubation, and length of intensive care unit stay.

DETAILED DESCRIPTION:
The patients will undergo the same preoperative preparation, intraoperative monitoring, and anesthetic technique. Fentanyl (2 μg/kg) will be given with induction of anesthesia, and additional increments of fentanyl 2 μg/kg will be administered if mean arterial blood pressure or heart rate rise in response to stressful surgical stimuli greater than 20% above baseline.

All surgeries will be performed through median sternotomy, with the same cardiopulmonary bypass and myocardial protection technique. At the end of surgery, all anesthetics will be discontinued, and patients will be transferred to the ICU where they will be committed to a mechanical ventilator.

the two blocks will be performed using Linear -Array ultrasound transducer probe (SONOSITE M-TURBO). After standard chest skin disinfection, the transducer will be covered with a sterile sleeve.

he two blocks will be performed using Linear -Array ultrasound transducer probe (SONOSITE M-TURBO). After standard chest skin disinfection, the transducer will be covered with a sterile sleeve.

Ultrasound guided Pecto-intercostal- fascial plane block:

The block will be performed while the patient in supine position after induction of general anesthesia and before skin incision. The probe of the ultrasound will be placed at 2 cm lateral to the lateral sternal border at 5th and 6th rib. On the surface plane subcutaneous tissue is identified, while Pectoralis major muscle, Intercostal muscles and ribs are seen in intermediate plane and lung along with pleura are identified in deep plane. A 22-gauge, 80-mm short bevel echogenic needle is used and advanced in in-plane manner, in a caudal-to-cranial direction, until the tip of the needle is located in the fascial plane between the pectoralis major and internal intercostal muscle, where the local anesthetic will be injected. As the drug will be injected, a hydro dissection of the plane is checked for. At this point, color doppler ultrasonography will be used to help identify the internal thoracic artery and its branches that pass through the plan.

Ultrasound guided erector spinae plane block:

The block will be done while the patient is in the sitting position before induction of general anesthesia. A high-frequency linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T6 spinous process corresponding to the T5 transverse process. Three muscles trapezius (uppermost), rhomboids major (middle), and erector spinae (lowermost) will be identified superior to the hyperechoic transverse process. Local infiltration with 2% of lignocaine at the site of needle insertion will be done. Using in-plane approach a 22 G short bevel needle will be inserted in caudal-cephalad direction, until the tip is deep to erector spinae muscle, as evidenced by visible hydro dissection below the muscle plane. A 20 ml of 0.25% plain bupivacaine will be injected on each side.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of either sex
* aged 18-50 years
* undergoing elective cardiac surgery via median sternotomy

Exclusion Criteria:

* refusal to participate,
* redo
* urgent cardiac surgery
* local infection of the skin at the site of needle puncture
* allergy to bupivacaine, coagulation disorders
* clinically significant liver or kidney disease, heart failure, moderate to severe pulmonary hypertension
* extubation is intentionally planned to be delayed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Total dose of fentanyl consumption | after 1 hour postoperative
  Analgesic effectiveness of both blocks in median sternotomy pain
Total dose of fentanyl consumption | after 24 hours postoperative
  Analgesic effectiveness of both blocks in median sternotomy pain

SECONDARY OUTCOMES:
time to extubation | after 1 hour of removal of endotracheal tube
  the time from ICU arrival till endotracheal extubation.
ICU Length of stay | after 48 hour postoperative
  length of intensive care unit stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Haasan Elhoshy, Alexandria, Egypt